CLINICAL TRIAL: NCT03039309
Title: Endoscopic Submucosal Dissection in the Treatment of Early Gastrointestinal Neoplasia: A UK Cohort Study to Assess Effectiveness and Safety
Brief Title: Endoscopic Submucosal Dissection for Early GI Neoplasia in the United Kingdom
Acronym: ESDUK
Status: Recruiting | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2016/45
Record Dates: First submitted 2017-01-23; First posted 2017-02-01 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Endoscopic Submucosal Dissection
Keywords: Endoscopic Submucosal Dissection
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection — Endoscopic submucosal dissection is an endoscopic resection technique that utilises an endoscopic knife to remove lesions within the gastrointestinal tract in an en bloc fashion.

SUMMARY:
Multicentre cohort study on the use of endoscopic submucosal dissection for the treatment of early gastrointestinal neoplasia.

DETAILED DESCRIPTION:
Data will be collected from participating centres on en bloc resection, curative resection, R0 resection and complications/adverse events over a 2 year follow up period.

Demographic details on the patients included in the study will be captured alongside details on the size and location of their early gastrointestinal dysplastic/neoplastic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above undergoing endoscopic submucosal dissection
* Participant is able to give informed consent for participation in the study

Exclusion Criteria:

* Patients under the age of 18
* Patients unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endoscopic submucosal dissection for early gastrointestinal neoplasia (e.g colorectal/gastric/oesophageal) in tertiary referral centres in the UK
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-08-05 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2028-08-04 (Estimated)

PRIMARY OUTCOMES:
Curative resection rate | 2 years
  % of successful resections free of disease at follow up endoscopy by the end of the follow up period (2 years)

SECONDARY OUTCOMES:
En bloc resection rate | At the time of procedure
  % of en bloc resections obtained at the time of initial endoscopic submucosal dissection
Complication rates | 28 days post procedure
  % of complications noted within 28 days following endoscopic submucosal dissection
Mortality rates | 2 years
  % of patients alive at the end of the 2 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Prof Pradeep Bhandari, MBBS, MD, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmputh Hospitals NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided